CLINICAL TRIAL: NCT06177041
Title: A Phase 3, Multi-Center, Double-Blind, Randomized, Efficacy and Safety Study of M108 Monoclonal Antibody Plus CAPOX Versus Placebo Plus CAPOX as First-line Treatment for Claudin (CLDN) 18.2-Positive, HER2-Negative, PD-L1 CPS<5, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma.
Brief Title: M108 Plus CAPOX Versus Placebo Plus CAPOX as First-line Treatment for Claudin (CLDN) 18.2-Positive, HER2-Negative, PD-L1 CPS<5, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: FutureGen Biopharmaceutical (Beijing) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FG-M108-04
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced Unresectable or Metastatic Gastric Cancer; Locally Advanced Unresectable or Metastatic Gastroesophageal Junction (GEJ) Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M108 plus CAPOX (Experimental)
  Interventions: Drug: M108 monoclonal antibody; Drug: Oxaliplatin; Drug: Capecitabine
- placebo plus CAPOX (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: M108 monoclonal antibody — M108 monoclonal antibody will be administered as a minimum 2-hour IV infusion.
  Arms: M108 plus CAPOX
Drug: Placebo — Placebo will be administered as a minimum 2-hour IV infusion.
  Arms: placebo plus CAPOX
Drug: Oxaliplatin — Oxaliplatin will be administered as a 2-hour IV infusion.
Drug: Capecitabine — Capecitabine will be administered orally twice daily (bid).

SUMMARY:
Gastric/GEJ adenocarcinoma, which is one of the major leading causes of cancer-related deaths worldwide, is a global challenge to human health. However, standard chemotherapy has limited efficacy in advanced gastric cancer, and there is an urgent need to explore and develop new therapeutic targets and combination therapy modalities. The main purpose of this study is to explore the efficacy of M108 monoclonal antibody plus capecitabine and oxaliplatin (CAPOX) versus placebo plus CAPOX as first-line treatment measured by progression free survival (PFS). This study will also evaluate safety, tolerability, pharmacokinetics and the immunogenicity profile of M108 monoclonal antibody, as well as its effects on quality of life.

DETAILED DESCRIPTION:
The aim of this phase 3, double-blind, randomized, placebo-controlled study is to explore the efficacy and safety of M108 monoclonal antibody plus chemotherapy versus placebo plus chemotherapy as first-line treatment for Claudin (CLDN) 18.2-Positive, HER2-Negative, PD-L1 CPS<5, locally advanced or metastatic gastric/GEJ adenocarcinoma. Patients will be randomized in a 1:1 ration to receive M108 monoclonal antibody plus chemotherapy or placebo plus chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Histologically confirmed diagnosis of locally advanced unresectable or metastatic gastric/GEJ adenocarcinoma with no treatment previously. For patients with neoadjuvant/adjuant chemotherapy in the past, duration of last therapy to recurrence should be more than 6 months
3. At least 1 measurable site of the disease according to RECIST 1.1 criteria.
4. Positive CDLN 18.2 expression
5. Negative HER2 expression, PD-L1 CPS<5
6. ECOG performance status (PS) 0-1
7. Life expectancy > 3 months
8. Age ≥ 18 years and ≤75 years
9. Adequate haematological/ coagulation/ hepatic/ renal function
10. Men and women of childbearing age should agree to use effective contraception from the time they sign their informed consent until 3 months after the last dosing. Female subjects of childbearing age must have a negative blood beta-HCG test within 72 hours prior to first dosing.

Exclusion Criteria:

1. Previous radiotherapy within 4 weeks prior to the start of study treatment. (if palliative radiotherapy was given to bone metastases and the patient recovered from acute toxicity was allowed).
2. Previous anti-tumor therapy within 4 weeks prior to the start of study treatment.
3. Previous major operation within 4 weeks prior to the start of study treatment.
4. Have a prior severe allergic reaction or intolerance to known components of M108 monoclonal antibodies or other monoclonal antibodies (including humanized or chimeric antibodies); Allergic or intolerant to any component of capecitabine, oxaliplatin, etc.
5. Subject who has been treated with CLDN18.2 monoclonal/bispecific antibodies, CLDN18.2 CAR-T, CLDN18.2 ADC and any therapies that target CLDN18.2.
6. Subject who is in pregnant or in lactation period.
7. Other clinically significant disease which may have adversely affected the safe delivery of treatment within this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2027-01-11 (Estimated); Study Completion 2027-04-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From date of randomization to the date of disease progression, death or end of study, assessed up to 24 months
  Compare PFS (Based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 by Independent Review Committee (IRC)) of patients treated with M108 monoclonal antibody or placebo plus CAPOX.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization to the date of death or end of study, assessed up to 24 months
  Compare OS (Based on RECIST 1.1 by IRC) of patients treated with M108 monoclonal antibody or placebo plus CAPOX.
Safety and tolerability assessed by adverse events (AEs) | From date of randomization until 28+7 days after the last dose
  An AE is any adverse medical event that occurs during a clinical study, whether or not related with medicinal product, including signs, symptoms, abnormal laboratory test results and diseases. The incidence and severity of AEs during the clinical study are recorded and analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China